CLINICAL TRIAL: NCT01315314
Title: Effects of Neutral pH and Low Glucose Degradation Product-containing Peritoneal Dialysis Fluid on Systemic Markers of Inflammation and Endothelial Dysfunction: a Randomized, Controlled 1-year Follow-up Study
Brief Title: Effect of Glucose Degradation Products (GDP) on Endothelial Dysfunction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kyungpook National University Hospital (Other)
Collaborators: Ministry of Health & Welfare, Korea (Other Government); Fresenius Medical Care Korea (Industry)
Responsible Party: Yong-Lim, Kim, Division of Nephrology and Department of Internal Medicine, Kyungpook National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IEDI MCS; A084001 (Other Grant/Funding Number: Ministry for Health and Welfare, Republic of Korea (A084001))
Record Dates: First submitted 2011-03-11; First posted 2011-03-15 (Estimated); Last update posted 2011-03-17 (Estimated); Status verified 2007-04

CONDITIONS: Kidney Failure, Chronic; Disorders Associated With Peritoneal Dialysis
Keywords: Glucose degradation products; Inflammation; Endothelial dysfunction; Soluble adhesion molecules; Peritoneal dialysis
MeSH Terms: conditions — Kidney Failure, Chronic; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- conventional PDF (Stay safe) (No Intervention)
- low GDP PDF (Balance) (Active Comparator)
  Interventions: Drug: Balance, Fresenius Medical Care, Germany

INTERVENTIONS:
Drug: Balance, Fresenius Medical Care, Germany — low glucose degradation product (GDP)-containing peritoneal dialysis fluid (PDF)
  Other Names: Balance, Fresenius Medical Care
  Arms: low GDP PDF (Balance)

SUMMARY:
The purpose of this study is to evaluate the effects of neutral pH and low glucose degradation product (GDP)-containing peritoneal dialysis fluid (PDF) on systemic inflammation and endothelial dysfunction markers in incident PD patients.

DETAILED DESCRIPTION:
New peritoneal dialysis fluids (PDF) with neutral pH and low glucose degradation products (GDPs) are used in patients on peritoneal dialysis (PD). Low GDP fluids are reported to be more biocompatible than conventional PDF. Determination of biocompatibility has mainly focused on local peritoneal effects; recently, there has been interest in evaluating the systemic biocompatibility of these fluids.

In recent analyses of two retrospective cohorts of Korean PD patients, significant survival advantage was shown for patients treated with the biocompatible PDF compared to patients treated with conventional PDF. However, the mechanisms of survival advantage with low GPD PDF in these observational studies are difficult to assess. Additionally, it is not clear that new PDFs favorably impact risk markers of cardiovascular disease (CVD).

Epidemiologic studies identified an independent association between inflammation and risk of cardiovascular events and mortality; this association has been confirmed in patients with advanced chronic kidney diseases (CKD).Other evidence showed that clinically overt vascular events are preceded by endothelial dysfunction and increases in circulating markers of endothelial activation, including vascular cellular adhesion molecule (VCAM)-1 and intercellular adhesion molecule (ICAM)-1.Moreover, there is an association between inflammation and elevated levels of soluble VCAM-1 and ICAM-1 in patients with or at risk of atherosclerosis. Elevated levels of soluble adhesion molecules are found in ESRD patients, especially in patients with CVD and malnutrition.

The investigators hypothesized that conventional PDF as well as uremia itself lead to local peritoneal changes such as peritoneal neoangiogenesis and fibrosis, effects related to ultrafiltration failure and subsequently volume overload. In addition, direct effect of GDPs and/or increased systemic levels of AGEs activate endothelial cells and increase levels of vascular adhesion molecules and inflammation. Both local and systemic effects of PDF are possibly associated with increased cardiovascular risks and mortality in PD patients.

This study aims to examine the effects of neutral pH and low GDP-containing PDF on systemic inflammation and endothelial dysfunction in incident PD patients in a randomized, controlled study.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged over 18 years and less than 75 years
* Within 90 days of initiation of first renal replacement treatment for ESRD
* Selected for maintenance management by CAPD
* Having provided informed consent
* Physically and mentally capable of performing the therapy

Exclusion Criteria:

* Patients were excluded if deemed to have less than 80% likelihood of survival for at least 1 year
* episodes of peritonitis within prior 30 days
* any malignancy other than treated skin carcinoma
* uncontrolled congestive heart failure
* recent (within 60 days) myocardial infarction or cerebrovascular accident
* active systemic vasculitic disease including systemic lupus erythematosus, polyarteritis nodosa, ANCA-nephritis, active rheumatoid disease, or active venous thrombotic-embolic disease
* any acute infection at the time of enrollment
* active or actively treated tuberculosis
* recent (within 30 days) systemic bacterial infection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2005-10; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Inflammation-endothelial-dysfunction index (IEDI) | Baseline and 12 months
  Inflammation-endothelial-dysfunction index (IEDI) is a composite score derived from measurement of serum levels of CRP (high sensitivity assay), soluble VCAM-1 and soluble ICAM-1. Changes between the groups will be tested by analysis of covariance (ANCOVA) with baseline values as covariates. Serial data will also be analyzed using a linear mixed model.

SECONDARY OUTCOMES:
Individual component markers of IEDI | Baseline and 12 months
  individual component markers of the IEDI including sICAM-1, sVCAM-1, and hs-CRP
RRF | Baseline and 12 months
  residual renal function (RRF) as average of urea and creatinine clearances by 24 hour urine collection
peritoneal clearance | Baseline and 12 months
  peritoneal clearance as weekly Kt/V urea and creatinine clearance
peritoneal ultrafiltration | Baseline and 12 months
  peritoneal ultrafiltration volume
peritoneal transport status | Baseline and 12 months
  dialysate-to-plasma ratio of creatinine at 4 hours of peritoneal equilibration test
serum albumin | Baseline and 12 months
LBM | Baseline and 12 months
  lean body mass (LBM) estimated from creatinine kinetics
nPNA | Baseline and 12 months
  normalized protein equivalent of nitrogen appearance (nPNA)
SGA | Baseline and 12 months
  subjective global assessment (SGA) with a four item and seven-point scale
Blood pressure | Baseline and 12 months
  systolic and diastolic blood pressure
use of antihypertensive medications | Baseline and 12 months
  number of antihypertensive medications
peritonitis rates | 12 months
  peritonitis rates
technique survival | 12months
  technique survival by Kaplan-Meier survival analysis with Log-Rank test.
patient survival | 12 months
  patient survival by Kaplan-Meier survival analysis with Log-Rank test.

CONTACTS AND LOCATIONS:
Overall Officials: Yong-Lim Kim, Professor, Study Chair — Kyungpook National University Hospital
Locations (1):
- Division of Nephrology and Department of Internal Medicine, Kyungpook National University Hospital, Daegu, South Korea